CLINICAL TRIAL: NCT00866463
Title: An Open-Label, Crossover Study In Healthy Volunteers To Evaluate The Pharmacokinetics Of Sildenafil Following Administration Of An Experimental Tablet Of Sildenafil With Or Without Water Relative To Viagra® Conventional Oral Tablet With Water.
Brief Title: A Study to Compare the Blood Levels of Sildenafil Following Administration of an Experimental Tablet vs. the Conventional Oral Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A1481265
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
Keywords: Sildenafil, Pharmacokinetics, Healthy Volunteer
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional Oral Tablet With Water (Active Comparator)
  Interventions: Drug: Sildenafil
- Experimental Tablet With Water (Experimental)
  Interventions: Drug: Sildenafil
- Experimental Tablet Without Water (Experimental)
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Single Dose of 50 mg Sildenafil Oral Tablet With Water
  Arms: Conventional Oral Tablet With Water
Drug: Sildenafil — Single Dose of 50 mg Sildenafil Experimental Tablet With Water
  Arms: Experimental Tablet With Water
Drug: Sildenafil — Single Dose of 50 mg Sildenafil Experimental Tablet Without Water
  Arms: Experimental Tablet Without Water

SUMMARY:
This study to will compare the blood levels of sildenafil following administration of an experimental tablet vs. the conventional oral tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between the ages of 18 and 55 years.
* Body Mass Index of 18 to 30 kg/m2, and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Smoking in excess of the equivalent of 5 cigarettes per day.
* Treatment with an experimental drug within 30 days or sildenafil, vardenafil, tadalfil within 4 days before first study dose.
* Develop blood pressure lowering or experience dizziness, lightheadedness when going from the laying down position to standing position.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Blood levels of sildenafil | 1 Day

SECONDARY OUTCOMES:
Blood levels of a metabolite of sildenafil | 1 Day
Side Effects | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481265&StudyName=A%20Study%20to%20Compare%20the%20Blood%20Levels%20of%20Sildenafil%20Following%20Administration%20of%20an%20Experimental%20Tablet%20vs.%20the%20Conventional%20Oral%20Tablet%20